CLINICAL TRIAL: NCT00399269
Title: Assessment of Efficacy & Safety of Recombinant Human Erythropoietin -Alpha, (rHu-EPO-Alpha) in Patients With Anemia of Chronic Renal Failure.
Brief Title: Efficacy & Safety Study of Recombinant Human Erythropoietin -Alpha, in Patients With Anemia of Chronic Renal Failure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cadila Pharnmaceuticals (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR - 50/9180
Record Dates: First submitted 2006-11-12; First posted 2006-11-14 (Estimated); Last update posted 2009-06-11 (Estimated); Status verified 2009-06

CONDITIONS: Anemia
Keywords: Anemia
MeSH Terms: conditions — Anemia

INTERVENTIONS:
Drug: Recombinant Human Erythropoietin alpha

SUMMARY:
To establish the efficacy and Safety of rHu-EPO-alpha in patients with anemia of Chronic Renal Failure.

DETAILED DESCRIPTION:
Despite impressive advances in the safety of the blood supply, the search for therapeutic alternatives to blood continues. Recombinant Human Erythropoietin (rHu-EPO), along with iron, vitamin B12, and folic acid, has been recommended as a specific medication that should be used instead of blood transfusion if the clinical condition of the patient permits sufficient time for these agents to promote erythropoiesis.

In normal physiological conditions Erythropoietin is produced in the kidney and stimulates the division and differentiation of committed erythroid progenitors in the bone marrow. rHu-EPO is a glycoprotein which stimulates red blood cell production. Epoetin alfa, a 165 amino acid glycoprotein manufactured by recombinant DNA technology, has the same biological effects as endogenous rHu-EPO.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 to 70 yrs of age of either sex.
* CRF patients who are EPO naïve or have been off EPO or similar Erythropoietic drugs for more than 4 weeks, falling with-in CKD stage III to V.
* Patients who are willing to give the consent
* Patient with Anemia of Chronic Renal Failure with Hb < 10.

Exclusion Criteria:

* Patients who are known hypersensitive to rHu-EPO.
* Patient's with history of anemia due to causes other than anemia of CRF.
* Patient's with history of Active infections, Hemoglobinopathies, Neoplastic diseases, and HIV infection.
* Patient's with history of G.I. bleeding (Overt or Occult).
* Patient's with history of serious or unstable medical or psychological conditions that could compromise the patient's safety or successful trial participation.
* Patients with abnormal liver function test. However, patients with HBsAg and HCV positive shall be included provided their Transaminases are normal.
* Female patient's of child bearing potential and not having undergone permanent sterilization procedures. Pregnant and lactating female patients.
* Patients unwilling or unable to comply with the study procedures. Chronic alcoholic or drug abuse patients

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2006-12; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Rise in Hemoglobin (Hb)/ Hematocrit (Hct) to therapeutic levels of 10 to 12 g/ dL
and/ or 30 to 36% respectively suggestive of normalized erythropoiesis at the end of study period of 12 Weeks.
OR
Rise in Hb by 1 g/ dL over two weeks of treatment with rHu-EPO.

SECONDARY OUTCOMES:
Rise of Hemoglobin and Haematocrit in CRF patients without significant adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. H. L. Trivedi, MD, Principal Investigator — IKDRC, Civil Hospital, Ahmedabad; Dr. Pankaj Shah, Nephrologist, Principal Investigator — IKDRC, Civil Hospital, Ahmedabad; Dr. Shishir Gang, Nephrologist, Principal Investigator — Muljibhai Patel Urological Hospital; Dr. Himanshu Patel, Nephrologist, Principal Investigator — Gujarat Kidney Foundation, Ahmedabad; Dr. Miten Mehta, Nephrologist, Principal Investigator — Anandabawa Kidney Dialysis Center, Jamnagar; Dr. Asit Mehta, Nephrologist, Principal Investigator — Apollo Hospitals, Ahmedabad
Locations (1):
- Dr. Shishir Gang, Nadiād, Gujarat, India